CLINICAL TRIAL: NCT07018037
Title: Pilot Study to Describe the Role of TTV During First-line Immunotherapy Treatment in Patients With Renal Cell Carcinoma
Brief Title: Role of TTV During First-line Immunotherapy Treatment in Patients With Renal Cell Carcinoma
Acronym: TTV ccRCC
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS289/IRE/25
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Renal Cell Carcinoma
Keywords: Torquetenovirus (TVV)
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this project is to descriptively explore the trend of torquetenovirus viral load TTV during therapy with immune checkpoint inhibitor ICI in these patients, to evaluate a possible role of this virus as a biomarker of response.

DETAILED DESCRIPTION:
The study involves the prospective recruitment of patients with metastatic clear cell renal cell carcinoma who begin a first line of treatment with immunotherapy at the UOC of Medical Oncology 1 of the Regina Elena Cancer Institute in Rome. Participants will undergo the following extra-clinical procedures and provided for by the protocol:

* Explanation, reading and signing of the informed consent;
* Performing a blood sample (approximately 7 ml);
* Collection of fecal material at different timepoints. It should be noted that the procedures necessary for conducting the study will not affect the diagnostic and therapeutic process of the patients and will only have research purposes.

The biological material collected, appropriately labeled, processed at the reference laboratories, where it will be used to perform the planned analyses. Blood and/or stool samples will be collected at different timepoints:

* Time zero (T0): before the start of therapy (blood and stool)
* C2 (T1): before the start of cycle 2 (blood)
* C4 (T2): after cycle 4, i.e. coinciding with the first radiological reassessment (blood and stool)
* 22W or 19W (T3): after 12 weeks from C4 i.e. coinciding with the radiological reassessments (blood and stool), i.e. at the last timepoint of this study.

Additional blood sampling will be performed in the case of immune-related toxicity (≥ G2 according to CTCAE) requiring steroid administration.

An additional sampling, as assessed by the investigating physician, will be collected at the time of disease progression (PD) (T4).

For each patient included in the study, the following data will be collected (obtained from the clinical documentation from the analyses conducted): personal/socio-demographic data (year of birth, sex, gender), complete histology and date of first diagnosis, surgical treatments, clinical data (e.g., laboratory tests), clinical data relating to the treatment (start and end date of each therapy with number of cycles administered, response to treatment, date of disease progression), date and location of each disease progression, patient status, date of last available follow-up, date of any death, data obtained from the analyses carried out within the present project.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age;
* Histological diagnosis of clear cell renal cell carcinoma;
* Evidence of advanced or metastatic disease;
* Patients diagnosed with metastatic clear cell renal cell carcinoma about to start first-line immunotherapy (ICI + ICI or ICI + TKI);
* Patients able to comply with the study procedures.
* Patients who give written informed consent personally or through a witness (study participation and data processing), before any study-specific procedure is started.

Exclusion Criteria:

* Previous neoplasms;
* Previous antineoplastic treatments;
* Previous steroid treatments;
* Active viral infections (e.g., HCV, HIV, etc.);
* Lack of autonomy in adhering to study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic clear cell renal cell carcinoma starting first-line immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Torquetenovirus in numbers of copies/ml | 24 months
  To descriptively evaluate the trend of torquetenovirus TTV viral load measured in number of copies/milliliter using a quantitative method, i.e. a REAL TIME PCR, during treatment with immunotherapy in patients with metastatic clear cell renal cell carcinoma starting a first-line treatment.

SECONDARY OUTCOMES:
Microbiome assessment | 24 months
  Microbiome will be described in terms of the type of microbial species present.

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy